CLINICAL TRIAL: NCT03324997
Title: Small Particle Hyaluronic Acid-Based Gel (Restylane Silk) for Treatment of Chest Wrinkles: A Randomized, Double-Blinded, Placebo-Controlled, Clinical Trial of Efficacy and Safety
Brief Title: Restylane Silk for Treatment of Chest Wrinkles
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Heidi Waldorf (Other)
Responsible Party: Sponsor-Investigator, Heidi Waldorf, Associate Clinical Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 16-2676
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Wrinkle
MeSH Terms: interventions — Sodium Chloride; Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Restylane (Experimental): half the chest to be treated with Restylane Silk
  Interventions: Drug: Restylane Silk; Device: Optical Coherence Tomography
- Placebo (Placebo Comparator): half-chest injections with saline as a placebo to Restylane Silk.
  Interventions: Drug: Saline; Device: Optical Coherence Tomography

INTERVENTIONS:
Drug: Restylane Silk — Restylane Silk is a temporary hyaluronic acid filler currently approved for the lips and fine lines around the mouth.
  Arms: Restylane
Drug: Saline — Saline as placebo
  Arms: Placebo
Device: Optical Coherence Tomography — An FDA-cleared non-invasive imaging device
  Other Names: OCT

SUMMARY:
The purpose of this study is to assess the safety and efficacy of using Restylane Silk to reduce the appearance of photoaging on the chest. Restylane Silk is a temporary hyaluronic acid filler currently approved for the lips and fine lines around the mouth. This study will compare the appearance of chest wrinkles on half the chest treated with Restylane Silk and the other half, which will be treated with placebo.

DETAILED DESCRIPTION:
Restylane Silk has been safely and effectively used in rejuvenation and appearance of wrinkles in the face. This study seeks to investigate the safety and efficacy of the injectable device in the chest for similar effects. Participants will undergo three treatments with Restylane Silk and results will be measured clinically and with Optical Coherence Tomography (an FDA-cleared non-invasive imaging device). Participants will receive randomized injections with the Restylane Silk product on half of the chest and will receive placebo injections on the other half. At the six-month period, participants will have the option to receive treatment with the product on the placebo side. At the 12-month period, participants may also elect for three additional touch-up treatments, which will not be counted as part of the study. If the chest is asymmetric in regards to wrinkles, the investigators will still proceed with the protocol because they are also comparing each side to itself prior to treatment, instead of simply comparing one side to the other.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 25-55 years.
* Moderate photodamaged skin of the chest/décolletage, as per the Fabi-Bolton chest wrinkle scale
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods and able to comply with all study requirements including daily applications of the study product, and restrictions regarding concomitant medication and other treatments.
* Female subject of childbearing potential must have a negative urine pregnancy test at screening and must be practicing an adequate, medically acceptable method of birth control for at least 30 days before Day 0 and at least 6 months after the last study product administration. Acceptable methods of birth control include intrauterine device (IUD); oral, transdermal, implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study); tubal ligation; abstinence and barrier methods with spermicide. Otherwise, if not of childbearing potential, subjects must: have a sterile or vasectomized partner; have had a hysterectomy, a bilateral oophorectomy or be clinically diagnosed infertile; or be in a menopausal state for at least a year.

Exclusion Criteria:

* History of keloid or hypertrophic scarring
* History of allergy or hypersensitivity to injectable hyaluronic acid gel, lidocaine, local topical anesthetics or nerve blocking agents
* Presence of any of the following at treatment sites: active inflammation/dermatitis, infection, psoriasis, herpes zoster, acanthosis, cancer, precancer, actinic keratosis
* History of the use of any other rejuvenate treatment in the preceding eight months or plans to use these substances or have these procedures during the study (including but not limited to neuromodulators, soft tissue augmentation, fractional resurfacing, chemical peel, ultrasound)
* The use of daily platelet inhibiting agents (i.e. Aspirin), anti-inflammatory medications, anticoagulants, Vitamin E, ginkgo biloba and other "herbs / homeopathic remedies" within 7 days of before or after treatment.
* History of severe allergies or multiple allergies manifested by Premarket Approval (PMA) P040024/s072: FDA Summary of Safety and Effectiveness Data page 10 anaphylaxis or a history of a hypotensive crisis in response to radio-contrast media or other osmotic agent
* Presence of any condition, which in the opinion of the investigator, would make the subject unable to complete the study per protocol
* Current use of immunosuppressive therapy
* History of connective tissue diseases such as rheumatoid arthritis, systemic lupus erythematous, polymyositis, dermatomyositis, or scleroderma;
* Participation in any interventional clinical research study within 30 days prior to randomization.
* Current smoker (or has quit smoking for less than 1 year)
* Current active malignancy

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-01-28 (Estimated); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Change in Fabi-Bolton (FB) clinometric chest wrinkle scale | Baseline and 6 months
  The change from baseline in blinded evaluator assessments of chest/décolletage and 6 months assessed by the Fabi-Bolton (FB) chest wrinkle. The Fabi-Bolton (F-B) 5-point wrinkle scale (1 = wrinkles absent; 2 = shallow but visible wrinkles; 3 = moderately deep wrinkles; 4 = deep wrinkles, with well-defined edges; 5 = wrinkles very deep with redundant folds).
Incidence of reported treatment emergent adverse events | up to 360 days
  The incidence of reported treatment emergent adverse events

SECONDARY OUTCOMES:
Change in dermal thickness | Baseline and 6 months
  Achieving statistically significant changes in optical coherence tomography (OCT) (epidermal, papillary, and visible reticular dermal thickness) at 6 months after 3 treatment sessions given
Change in papillary dermal brightness | Baseline and 6 months
  Achieving statistically significant changes in OCT parameters (papillary dermal brightness) at day 180 after 3 treatment sessions given
Change in upper dermal reflectivity | Baseline and 6 months
  Achieving statistically significant changes in OCT parameters (upper dermal reflectivity) at day 180 after 3 treatment sessions given
Change in dermoepidermal contrast | Baseline and 6 months
  Achieving statistically significant changes in OCT parameters (dermoepidermal contrast) at day 180 after 3 treatment sessions given
Change in surface contouring | Baseline and 6 months
  Achieving statistically significant changes in OCT parameters (surface contouring) at day 180 after 3 treatment sessions given
Patient satisfaction | 6 months
  The questionnaire consists of two "Yes/No" questions (score 0 or 1) and five questions using a 5 point Likert rating scale with scores ranging from 0 (extremely dissatisfied) to 5 (extremely satisfied). The total score range is from 0-27.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Waldorf, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Giselle Singer, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States